CLINICAL TRIAL: NCT00361556
Title: Treatment for Nonspecific Low Back Pain in Primary Care With Standardized Health Education Booklets: A Randomized Controlled Clinical Trial
Brief Title: Treatment for Nonspecific Low Back Pain in Primary Care: a Trial on Different Health Education Booklets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Collaborators: Spanish Back Pain Research Network (REIDE) (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Carmen Fernández, Centro de Salud de Valldargent, Kovacs Foundation
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FK-R-11
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Low Back Pain
Keywords: low back pain; disability; health education; primary care
MeSH Terms: conditions — Low Back Pain; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): The Back Book
  Interventions: Behavioral: The Back Book; Behavioral: The Back Guide; Behavioral: General health book
- 2 (Active Comparator): The Back Guide
  Interventions: Behavioral: The Back Guide; Behavioral: General health book
- 3 (Active Comparator): General health book
  Interventions: Behavioral: General health book

INTERVENTIONS:
Behavioral: The Back Book — A book on how to prevent back pain
  Arms: 1
Behavioral: The Back Guide — A guide for the prevention of back pain.
  Arms: 1; 2
Behavioral: General health book — A book on general health

SUMMARY:
The primary purpose of this study is to compare the effectiveness on the disability of low back pain patients of The Back Book, The Back Guide, and a control intervention (generic recommendations on general health). Patients are divided into 3 groups:those who receive The Back Book (classic education), those who receive The Back Guide (cognitive behavioral education) and the control group). They are patients who consult a physician at the primary care consults of 14 different Health Centers in Spain. The sample size is 240 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain patients,
* with or without referred or radiated pain;
* without red flags for systemic disease or criteria for surgery.

Exclusion Criteria:

* Inability to read the handout or to fill out the questionnaires;
* habitually in a prostrate position;
* diagnosis of inflammatory rheumatologic disease, cancer or fibromyalgia; suspicion of fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-10; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Degree of disability at 180 days of follow-up. | 6 months

SECONDARY OUTCOMES:
Catastrophizing and days on sick leave at 180 days of follow-up. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M. Kovacs, MD, PhD, Study Chair — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Carmen Fernández, MD, Principal Investigator — Centro de Salut de Valldargent, Palma de Mallorca 07013, Spain; Antonio Ruiz, MD, Study Director — Centro de Salud Las Ciudades, Madrid 28903, Spain; Carlos Isanta, MD, Study Director — Centro de Salud de San José, Zaragoza 50013, Spain; Violeta González, MD, Study Director — Centro de Salud Gazteleku, Bilbao 48007, Spain; Pablo Panero, MD, Study Director — Centro de Salud de Órgiva, Órgiva, Granada 18400, Spain; Margarita Gómez, MD, Study Director — Centro de Salud Casa del Mar, Palma de Mallorca 07012, Spain; Francisco Martínez, MD, Study Director — Centro de Salud de Bembibre, Bembibre, León 24300, Spain; Luis González, MD, Study Director — Centro de Salud Serrería II, Valencia 46022, Spain; Sergio Giménez, MD, Study Director — Centro de Salud de Ciudad Jardín, Málaga 29017, Spain
Locations (1):
- Primary care Centers affiliated with the Spanish Back Pain Research Network, Throughout Spain, Spain

REFERENCES:
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Cherkin DC, Eisenberg D, Sherman KJ, Barlow W, Kaptchuk TJ, Street J, Deyo RA. Randomized trial comparing traditional Chinese medical acupuncture, therapeutic massage, and self-care education for chronic low back pain. Arch Intern Med. 2001 Apr 23;161(8):1081-8. doi: 10.1001/archinte.161.8.1081. PMID 11322842
- [Background] Hagen EM, Eriksen HR, Ursin H. Does early intervention with a light mobilization program reduce long-term sick leave for low back pain? Spine (Phila Pa 1976). 2000 Aug 1;25(15):1973-6. doi: 10.1097/00007632-200008010-00017. PMID 10908942
- See also: Spanish Back Pain Research Network site that describes objectives and projects of its members. — http://www.reide.org